CLINICAL TRIAL: NCT00193739
Title: A Prospective Randomized Trial of Neoadjuvant Chemotherapy and Surgery Versus Concurrent Chemoradiation Therapy in Patients With Stage IB2-IIB Squamous Carcinoma of the Uterine Cervix
Brief Title: Neoadjuvant Chemotherapy Followed by Surgery Versus Concurrent Chemoradiation in Carcinoma of the Cervix
Acronym: NACTcervix
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Tata Memorial Hospital (Other Government)
Responsible Party: Principal Investigator, Sudeep Gupta, Professor of Medical Oncology, Tata Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 119 of 2003
Record Dates: First submitted 2005-09-11; First posted 2005-09-19 (Estimated); Last update posted 2019-09-20 (Actual); Status verified 2019-09

CONDITIONS: Cancer of Cervix
Keywords: Neoadjuvant chemotherapy; Surgery; Cervix cancer; Concurrent chemoradiation
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Neoadjuvant Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- NACT followed by surgery (Active Comparator): 3 cycles of neoadjuvant chemotherapy (NACT) (Inj.Paclitaxel +Inj.Carboplatin) followed by surgery (radical abdominal hysterectomy Class III , bilateral pelvic lymphadenectomy & lower para aortic lymph node sampling)
  Interventions: Drug: NACT; Procedure: Radical abdominal hysterectomy (class III), BPLND & lower para aortic lymph node sampling
- Concurrent chemoradiotherapy (Active Comparator): Radiation therapy will be administered to whole pelvis followed by intracavitary brachytherapy. Patients will be given chemotherapy (Inj.Cisplatin) concurrently with external beam radiotherapy.
  Interventions: Drug: Inj.Cisplatin; Radiation: Concurrent chemo radiotherapy

INTERVENTIONS:
Drug: NACT — 3 cycles of neoadjuvant chemotherapy
  Other Names: Neoadjuvant chemotherapy (Inj.Paclitaxel + Inj.Carboplatin)
  Arms: NACT followed by surgery
Procedure: Radical abdominal hysterectomy (class III), BPLND & lower para aortic lymph node sampling — NACT followed by surgery
  Other Names: Radical abdominal hysterectomy (class III), bilateral pelvic lymphadenectomy & lower para aortic lymph node sampling
  Arms: NACT followed by surgery
Drug: Inj.Cisplatin — Concurrent chemo radiotherapy
  Arms: Concurrent chemoradiotherapy
Radiation: Concurrent chemo radiotherapy — Radiation therapy will be administered to the whole pelvis region followed by intracavitary brachytherapy.
  Other Names: External beam radiotherapy followed by intracavitary brachytherapy. (EBRT + ICA)
  Arms: Concurrent chemoradiotherapy

SUMMARY:
Carcinoma cervix is a common malignancy in women in developing countries including India. The standard treatment of locally advanced cervical cancer (Stages IB2 to IIIB)is concomitant chemoradiation (CT RT) using platinum based chemotherapy. Some studies, including a meta-analysis conducted by the Cochrane group, have indicated that few courses of neoadjuvant chemotherapy (NACT) followed by surgery may be superior to radical radiation alone for these patients. However NACT-Surgery approach has never been compared to the current standard of concomitant CT RT. The present study is undertaken to compare, in a randomized trial, NACT(3 courses of paclitaxel-carboplatin) followed by surgery to concomitant CT RT in stages IB2 to IIB squamous cell carcinoma of the uterine cervix.

DETAILED DESCRIPTION:
Cancer of the uterine cervix is a major health problem in the developing countries including India and is the commonest cancer amongst women in India with nearly 1,00000 new women diagnosed to have this cancer every year. It is also the main cause of cancer related mortality among women in India. At the Tata Memorial Hospital, approximately 1600 new patients with cervical cancer are registered every year, of which nearly 70% present in locally advanced stages.

A majority of patients diagnosed with stage IB cervical cancer in India have bulky tumours (more than 4 cm in size) and have now been classified as stage IB2 as per the new FIGO staging (1). These tumours are associated with a high incidence of pelvic lymph node metastases. Finan et al (2) noted positive pelvic nodes in 15.5% of patients with stage Ib1 disease versus 43.8% with stage Ib2. Positive paraaortic nodes were present in 1.8% of patients for stage Ib1 disease versus 6.3% of patients with stage Ib2. The result of radical surgery and radical radiation therapy alone or in combination in these tumours has been reported to be much inferior to stage IB1 tumours (60-65% vs. 85-90% five year survival). The incidence of pelvic lymph node metastasis and the results of treatment of stage IB2 tumours are more or less similar to those with stage IIB tumours.

The ability of radiotherapy or surgery to cure locally advanced cervical cancer is limited by the size of the tumour, high incidence of pelvic lymph node metastases and potential for systemic spread. Besides, the doses required to treat large tumours exceed the limit of toxicity in normal tissue. Efforts to overcome this problem have included the use of different chemotherapy drugs in different schedules. Chemotherapy has been used in the management of locally advanced cervical cancers along with radiation therapy and surgery in different ways e.g. neoadjuvant, adjuvant and concurrent.

The standard approach to using chemotherapy in the treatment of patients with locally advanced disease is the use of concurrent chemoradiation. The concurrent use of single drug and multiple drug regimens with radiotherapy has been tested in women with cervical cancer. Recent data from prospective randomised trials and two meta-analyses (3-12) has unequivocally shown significant survival advantage (both disease free and overall survival) with the use of concurrent chemoradiation using platinum based chemotherapy compared to radical radiation alone in patients with locally advanced cervical cancer (stages IB2-IIIB). A significant reduction in distant metastases was also noted in the concurrent chemoradiation therapy arm. This has led to acceptance of concurrent chemoradiation therapy as the new standard of care for locally advanced cervical cancer. The meta-analyses of these trials showed that the beneficial effect on survival was more evident in stage IB2 and stage II B tumours compared to stage III B tumours (which constituted only about 35% of total number of patients).

An alternative approach is to use chemotherapy prior to local therapy, which could be surgery or radiation. Some theoretical benefits of neoadjuvant chemotherapy (hereinafter abbreviated as NACT) like eradication of micrometastases have long been advanced but never proven. It certainly helps in the reduction of tumour bulk in some patients with locally advanced disease. Some of these latter patients are then able to undergo surgery which is otherwise not possible. The downside to NACT is the delay in institution of definitive treatment in the 20 to 30% patients who don't respond to chemotherapy. The randomized trials of NACT followed by radiation therapy versus radiation therapy alone showed no improvement in survival (13-19). It is possible that the failure to show a survival benefit with NACT followed by radiation is due to the selection of chemoresistant clones which are also radioresistant. A second explanation (also advanced for the failure of NACT approach in head and neck cancers) is that NACT just selects out the patients (the ones who respond) who have biologically favourable disease and confers no benefit by itself. Surgical removal of the tumour after chemotherapy will however have no interaction with biochemical resistance of the remaining clones. It therefore has the potential of providing a benefit additive to chemotherapy and radiotherapy. In their papers Sardi et al (20, 21) reported on their randomized trial of NACT (bleomycin, vincristine and cisplatin) followed by surgery plus radiation versus either surgery plus radiation or radiation as the control arm in patients with stage 1B, 2B and 3B cervical cancer. There was a high response rate to NACT in stage 1B patients (90% in 1B1 and 83.6% in 1B2). The overall survival in the whole group of stage 1B patients was superior in the NACT arm (n=102) compared to the control arm (n=103) (81% Vs 66%, p = 0.025). The resectability rate among stage 1B2 patients given NACT was 100% (n = 61) compared to 85% in the controls (n = 56). In stage 2B the resectability rate in the NACT arm was 80% (n = 76) compared to 56% in the control arm (n = 75). However there was no clear survival advantage of the NACT arm over controls in stages 2B and 3B. Although this trial has reported a survival advantage of NACT followed by surgery in a subgroup of patients its results are not definitive. The treatment offered in the control arm of this trial (attempt at surgical removal upfront in stages 1B and 2B or radiation only in stages 2B and 3B) was not standard by current standard and the numbers in various groups were small. In order to be considered a therapeutic option in locally advanced patients, NACT followed by surgery must be compared to the current therapeutic standard, which is concurrent chemoradiation. The chemotherapeutic options for cervical cancer at present are different from the one used by Sardi et al. The combination of ifosfamide and cisplatin or paclitaxel and carboplatin is likely to show a higher response rate compared to the regimen used by Sardi et al, which was bleomycin, vincristine and cisplatin.

Considering these results from the literature, it appears logical to compare neoadjuvant chemotherapy followed by surgery with concurrent chemoradiation in patients with stage IB2 to IIB squamous carcinoma of the cervix.

ELIGIBILITY:
Inclusion Criteria:

1. Women with histologically proven invasive squamous cell carcinoma of the uterine cervix, stages IB2-IIB.
2. Age 18-65 years (both inclusive)
3. No evidence of visceral, skeletal or extra-abdominal nodal metastases.
4. No history of prior or present second malignancy
5. Good performance status (Karnofsky performance score > 70 or ECOG PS <2)
6. Normal hematological & biochemical parameters including normal renal function.
7. Presence of associated co-morbid conditions that preclude participation in the study.
8. No prior treatment.
9. Informed consent for participation in the study.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 635 (Actual)
Dates: Start 2003-09-04 (Actual); Primary Completion 2020-07-31 (Estimated); Study Completion 2020-07-31 (Estimated)

PRIMARY OUTCOMES:
Disease Free Survival | 5 years
  Disease free survival will be calculated from the date of entry into the study to the date of first physical or radiographic evidence disease relapse or death due to disease or last follow up visit.

SECONDARY OUTCOMES:
Over all survival | 7 years
  Over all survival will be calculated from the date of entry into the study to the date of death due to any cause or the last follow up visit.
Rate of Distant Metastases | 7 years

CONTACTS AND LOCATIONS:
Overall Officials: Sudeep Gupta, MD, DM, Principal Investigator — Tata Memorial Hospital, Mumbai-400012,India; Shyam K Shrivastava, MD, Principal Investigator — Tata Memorial Hospital, Mumbai-400012, India
Locations (1):
- Tata Memorial Hospital, Mumbai, Maharashtra, India

REFERENCES:
- [Result] 928O_PRNeoadjuvant chemotherapy followed by surgery (NACT-surgery) versus concurrent cisplatin and radiation therapy (CTRT) in patients with stage IB2 to IIB squamous carcinoma of cervix: A randomized controlled trial (RCT) S. Gupta P. Parab R. Kerkar U. Mahantshetty A. Maheshwari S. SastriR. Engineer R. Hawaldar J. Ghosh S. Gulia ... Show more Annals of Oncology, Volume 28, Issue suppl_5, 1 September 2017, mdx440.038,https://doi.org/10.1093/annonc/mdx440.038 Published: 18 September 2017
- [Result] Gupta S, Maheshwari A, Parab P, Mahantshetty U, Hawaldar R, Sastri Chopra S, Kerkar R, Engineer R, Tongaonkar H, Ghosh J, Gulia S, Kumar N, Shylasree TS, Gawade R, Kembhavi Y, Gaikar M, Menon S, Thakur M, Shrivastava S, Badwe R. Neoadjuvant Chemotherapy Followed by Radical Surgery Versus Concomitant Chemotherapy and Radiotherapy in Patients With Stage IB2, IIA, or IIB Squamous Cervical Cancer: A Randomized Controlled Trial. J Clin Oncol. 2018 Jun 1;36(16):1548-1555. doi: 10.1200/JCO.2017.75.9985. Epub 2018 Feb 12. PMID 29432076